CLINICAL TRIAL: NCT02066896
Title: Low Level Laser Therapy For The Treatment Of Xerostomia In Primary Sjogren's Syndrome
Brief Title: Laser Therapy to Treat the Dry Mouth of Sjogren's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, TANIA SALES DE ALENCAR FIDELIX, DR., Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLLXS
Record Dates: First submitted 2013-08-15; First posted 2014-02-20 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-04

CONDITIONS: KERATOCONJUNCTIVITIS SICCA; XEROSTOMIA; SICCA SYNDROME; PRIMARY SJOGREN SYNDROME
Keywords: Sjogrens Syndrome; Syndrome, Sjogren's; Sjogren Syndrome; Sicca Syndrome; Syndrome, Sicca
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Xerostomia; Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Comparator: Sham Lasertherapy (Sham Comparator): Sham lasertherapy in parotid, submandibular and sublingual glands for six weeks.
  Interventions: Device: Sham Lasertherapy
- Active Comparator: Lasertherapy (Active Comparator): Low level lasertherapy in parotid, submandibular and sublingual glands for six weeks.
  Interventions: Device: Lasertherapy

INTERVENTIONS:
Device: Lasertherapy — Laser 808 wave length infrared Ga AlAs(gallium-aluminum-arsenide). The laser beam applied bilaterally in non contact mode to each salivary gland area, extra orally to the parotid and submandibular glands and intramurally to the sublingual gland/ 4 Joules/cm2 each point (active group)
  Arms: Active Comparator: Lasertherapy
Device: Sham Lasertherapy — Laser 808 wave length infrared Ga AlAs(gallium-aluminum-arsenide).The device will be applied with the laser pen closed by aluminium foil (placebo group).
  Arms: Sham Comparator: Sham Lasertherapy

SUMMARY:
This study was designed to test the efficacy and safety of low laser therapy to treat the xerostomia of patients with primary Sjogren's Syndrome.

DETAILED DESCRIPTION:
The Sjogren's Syndrome is a disease that affects around 0,5% of the population and is mainly characterized for inflammatory involvement of salivary and lacrimal glands.

The xerostomia leads to low quality of life caused by dry sensations that can disturb the taste, the speaking, the swallow and chewing functions in the affected patients. The absent saliva can cause increase of dental caries and decays.

Until now, there is no effective treatment that increases the amount of saliva and the patients have low improvements with cholinergic drugs such as pilocarpine and cevimeline. These drugs can cause unpleasant collateral effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary Sjogren Syndrome according criteria american european 2002.
* Salivary flux non stimulated < 0,1 ml/min.

Exclusion Criteria:

* hepatitis B and/or C
* radiotherapy in the glandular area (previous)
* other connective diseases
* thyroidopathy non compensated
* GVHD graft-versus-host disease
* HIV
* Sarcoidosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia M Trevisani, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Tania S A Fidelix, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fidelix T, Czapkowski A, Azjen S, Andriolo A, Neto PH, Trevisani V. Low-level laser therapy for xerostomia in primary Sjogren's syndrome: a randomized trial. Clin Rheumatol. 2018 Mar;37(3):729-736. doi: 10.1007/s10067-017-3898-9. Epub 2017 Nov 9. PMID 29119483

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study sample consisted of 66 patients who were selected from 84 patients referred from ophthalmology and rheumatology division of university hospital. The patients met primary Sjögren's criteria (2002).
Pre-assignment Details: The exclusion criteria were: sarcoidosis, uncontrolled thyroidopathy, HIV and HCV infections and head or neck irradiation history. A computer-generated randomization list was used to allocate patients ramdomly into two groups: active laser therapy and sham laser therapy. Concealed randomization was performed with opaque sealed envelopes.
Period: Overall Study
Arm/Group | Sham Comparator: Sham Lasertherapy | Active Comparator: Lasertherapy
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Comparator: Sham Lasertherapy | Active Comparator: Lasertherapy | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Median (Standard Deviation); unit: years (SD)] | 58 (11.1) | 54 (11.3) | 57 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: The Xerostomia Inventory
Description: The Xerostomia Inventory (XI) is an 11-item questionnaire (Thomson et al, 1999). Scores to the 11 items are summated, providing a single score (5-55) representing the subjective severity of xerostomia. In 2012, da Mata published a validated version in portuguese and we used this version. The better score is the lowest. The significant variation is defined as 6 or more.
  Bellow we describe all the 11 questions:
  1. I sip liquids to aid in swallowing food
  2. My mouth feels dry when eating a meal
  3. I get up at night to drink
  4. My mouth feels dry
  5. I have difficulty in eating dry foods
  6. I suck sweets or cough lollies to relieve dry mouth
  7. I have difficulties swallowing certain foods
  8. The skin of my face feels dry
  9. My eyes feel dry
  10. My lips feel dry
  11. The inside of my nose feels dry __________________________________________________________
  Score:
  Never' (1), Hardly ever' (2), Occasionally' (3), Fairly often' (4), Very often' (5)
Time Frame: 6 weeks
Population: Intent to treat population. Last observation carried forward imputation method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Comparator: Sham Lasertherapy | Active Comparator: Lasertherapy
Number analyzed (Participants) | 33 | 33
units on a scale | 40.2 (8.3) | 39.3 (8.1)
Statistical Analysis 1: Comparison: Sham Comparator: Sham Lasertherapy vs Active Comparator: Lasertherapy; Test type: Other — ANOVA repeated measures; p = 0.05, ANOVA; ANOVA repeated measures

2. Secondary Outcome: Salivary Biomarker Analysis. Beta 2 Microglobulin.
Description: The saliva in Sögren's syndrome patients has a high level of beta 2 microglobulin reflecting progression of the disease and inflammatory process at glandular epithelium.
  The saliva samples were collected at the baseline and end point. Beta 2 microglobulin was determined by Elisa human kit (ABCAM ab 108885).
  The normal levels are 1,2 +/- 0,7 microg/ml, and for primary Sjögren's syndrome 5,3 +/- 4,6 microg/ml.
  This measure was done in the samples of saliva before and after the lasertherapy for all patients.
Time Frame: 6 weeks
Measure: Median (Standard Deviation); unit: microg/ml
Arm/Group | Sham Comparator: Sham Lasertherapy | Active Comparator: Lasertherapy
Number analyzed (Participants) | 33 | 33
microg/ml | 1.10 (3.63) | 0.84 (4.93)

3. Secondary Outcome: Salivary Flux Measurement
Description: The salivary flux was measured at the same time, without previous meal or tooth brushing, drinking or eating, in a quiet room. Spilled saliva was collected in a graduated Falcon 15ml tube. The samples of saliva were frozen and stored at -20° C.
  Normal salivary stimulated flux is above 0,5 ml/min. Normal unstimulated salivary flux is above 0,2 ml/min.
Time Frame: 6 weeks
Measure: Median (Standard Deviation); unit: ml/min
Arm/Group | Sham Comparator: Sham Lasertherapy | Active Comparator: Lasertherapy
Number analyzed (Participants) | 33 | 33
ml/min | 0.100 (0.164) | 0.100 (0.114)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Sham Comparator: Sham Lasertherapy | Active Comparator: Lasertherapy
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No